CLINICAL TRIAL: NCT02098655
Title: Analysis of the Parameters Obtained on Stabilometric Platform in Patients With Parkinson's Disease: a Basis for a Rehabilitation Perspective
Brief Title: Analysis of the Parameters Obtained on Stabilometric Platform in Patients With PD
Acronym: SPPD001
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: SP PD 001; SP PD 001 (Other: Ospedale Generale di Zona Moriggia-Pelascini)
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson's Disease; Disturbance; Balance, Labyrinth; Other Falls
Keywords: Stabilometric Platform; Postural instability
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 30 patients with PD: 30 patients (12 M, 18 F, mean age 66,8 ± 8,7) with PD in stage 3 of H&Y will undergo training of balance using a stabilometric platform
  Interventions: Other: Stabilometric platform
- 12 healthy volunteers: 12 healthy volunteers (3 M, 9 F, mean age 66,5 ± 6,0) served as controls will undergo training of balance using a stabilometric platform
  Interventions: Other: Stabilometric platform

INTERVENTIONS:
Other: Stabilometric platform — Stabilometric platform is a device used for assessment and training of balance basing on ground reaction force evaluation in static conditions.

SUMMARY:
Objective: To analyze different parameters in patients with Parkinson's Disease (PD) obtained through the use of a stabilometric platform and compare them with those of a control population. To interpret the data in order to find some postural instability indicators that can become useful to build a rehabilitation strategy for balance disorders in PD.

DETAILED DESCRIPTION:
Background: Posture and balance are the foundation on wich upright stance and walking are executed. Postural instability is the impairment in balance that compromises the ability to maintain or change posture such as standing and walking. It is considered to be one of the cardinal features of PD. In such patients it is present even at diagnosis and worsens with disease progression. It correlates with falls representing a major source of disability and reduced QoL in PD. In this course, the study of balance is important to identify patients who can benefit from specific rehabilitative treatment.

Objective: To analyze different parameters in patients with PD obtained through the use of a stabilometric platform and compare them with those of a control population. To interpret the data in order to find some postural instability indicators that can become useful to build a rehabilitation strategy for balance disorders in PD.

ELIGIBILITY:
Inclusion Criteria:

* PD according to Gelb et al., in Hoehn-Yahr stage 3, with the ability to walk without any assistance, who had fallen in the last year at least 2 times, with mini-mental state examination score ≥26.
* Healthy volunteers

Exclusion Criteria:

* atypical parkinsonism
* patients with cerebro-vascular disorders or other neurological conditions including cognitive impairment.
* patients with relevant comorbidity or vestibular/visual dysfunctions limiting locomotion or balance.

Ages: 58 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Trunk sway | One week
  With respect to the average centre of gravity the Standard Deviation of trunk sway (total, in Antero-Posterior and in Medio-Lateral direction) were calculated. In this way it was possible to obtain a statokinesigram, that is the layout of a line connecting the successive positions of the center of pressure during the recording, and the area of the ellipse containing 90% of the sampled positions of the center of pressure. These measurements were obtained with open eyes (OE), and while the patient performing a cognitive task (counting).

SECONDARY OUTCOMES:
BBS | One week
  Berg Balance Scale

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Parkinson disease and movement disorders rehabilitation unit, Ospedale Generale di Zona "Moriggia-Pelascini", Gravedona ed Uniti (CO), Italy
Locations (1):
- Ospedale Generale di Zona "Moriggia-Pelascini", Gravedona, Como, Italy